CLINICAL TRIAL: NCT06304324
Title: Perineural Dexmedetomidine Vs Dexamethasone on the Duration of Popliteal Nerve Block for Anesthesia After Pediatric Ankle Surgery
Brief Title: Dexmedetomidine Vs Dexamethasone in Popliteal Nerve Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18/2023
Record Dates: First submitted 2024-01-22; First posted 2024-03-12 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-01

CONDITIONS: Ankle Disease; Ankle Injuries and Disorders; Foot Injury; Foot Diseases
MeSH Terms: conditions — Ankle Injuries; Disease; Foot Injuries; Foot Diseases | interventions — Sodium Chloride; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sham Block (Placebo Comparator): 0.2% ropivacaine for popliteal nerve block
  Interventions: Drug: 0.9% Sodium chloride
- Dexamethasone (Active Comparator): 0.1mg/kg dexamethasone added to 0.2% ropivacaine for popliteal nerve block
  Interventions: Drug: 0.1mg/kg Dexamethasone
- Dexmedetomidine (Active Comparator): 0.5ug/kg dexmedetomidine added to 0.2% ropivacaine for popliteal nerve block
  Interventions: Drug: 0.05ug/kg Dexmedetomidine

INTERVENTIONS:
Drug: 0.9% Sodium chloride — administration of 0.5ml/kg of 0,2% ropivacaine + 0.01ml/kg 0.9% sodium chloride for the popliteal nerve block
  Other Names: placebo
  Arms: Sham Block
Drug: 0.1mg/kg Dexamethasone — administration of 0.5ml/kg of 0.2% ropivacaine with 0.1mg/kg Dexamethasone for the popliteal nerve block
  Arms: Dexamethasone
Drug: 0.05ug/kg Dexmedetomidine — administration of 0.5ml/kg of 0.2% ropivacaine with 0.05ug/kg dexmedetomidine for the popliteal nerve block
  Arms: Dexmedetomidine

SUMMARY:
Effect of Perineural Dexmedetomidine vs. Dexamethasone on the duration of popliteal nerve block for Anesthesia After Pediatric ankle/foot surgery.

DETAILED DESCRIPTION:
This study is proposed to explore the effect of systemic Dexamethasone on the duration of popliteal block for analgesia after pediatric ankle surgery.

After ankle/foot surgery, children need good analgesia. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe.

The safety of local anaesthesia is essential in children due to the much lower toxicity threshold of local anaesthetics. An effective adjuvant, such as Dexamethasone, could allow for a higher dilution of local anaesthetics while maintaining and enhancing their analgesic effect.

There is considerable research where intravenous and perineural dexamethasone use has been compared in adults. However, there is a massive lack of research regarding children.

In this study, investigators compare perineural Dexmedetomidine and Dexamethasone. Group 2 will have Dexamethasone in a 0.1mg/kg dose, and group 2 will have dexmedetomidine in a 0.5 ug/kg dose added to the local anaesthetic in peripheral nerve block.

The investigator's goal is to find which perineural adjuvant, Dexamethasone or dexmedetomidine, covers the need for good pain relief and fast recovery postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* children scheduled for foot/ankle surgery
* body weight > 5kg

Exclusion Criteria:

* infection at the site of the regional blockade
* coagulation disorders
* immunodeficiency
* ASA= or >4
* steroid medication in regular use

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
time to the first need of opiate following the procedure | within 48 hours
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale | 4 hours
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain in individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale | 6 hours
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain in individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale | 8 hours
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain in individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale | 12 hours
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain in individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale | 16 hours
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain in individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale | 20 hours
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain in individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale | 24 hours
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain in individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale | 36 hours
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain in individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale | 48 hours
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain in individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Neutrophil-to-lymphocyte ratio | 24 hours after surgery
  Neutrophil to lymphocyte ratio (NLR) is used as a marker of subclinical inflammation. It is calculated by dividing the number of neutrophils by number of lymphocytes, usually from peripheral blood sample.
Platelet-to-lymphocyte ratio | 48 hours after surgery
  The platelet-lymphocyte ratio (PLR) is a novel inflammatory marker, which may be used in many diseases for predicting inflammation and mortality. The PLR can be easily calculated and is widely available but it may be affected by several inflammatory conditions.
Platelet-to-lymphocyte ratio | 24 hours after surgery
  The platelet-lymphocyte ratio (PLR) is a novel inflammatory marker, which may be used in many diseases for predicting inflammation and mortality. The PLR can be easily calculated and is widely available but it may be affected by several inflammatory conditions.
Time to mobilization | within 48 hours
  Time after surgery when the patient moves the toe for the first time

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Kotwicki, Prof dr hab, Study Chair — Poznan University of Medical Sciences
Locations (1):
- Department of Spine Diseases and Pediatric Orthopedics, University of Medical Sciences, Poznań, Poland, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No